CLINICAL TRIAL: NCT00081406
Title: Child and Family Therapy for Anxiety-Disordered Youth
Brief Title: Individual and Family Therapy for Children With Anxiety Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH059087 (NIH); R01MH059087 (NIH); DSIR CT-S
Record Dates: First submitted 2004-04-09; First posted 2004-04-12 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2005-03

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Educational Status

INTERVENTIONS:
Behavioral: Individual Child CBT
Behavioral: Family CBT
Behavioral: Education/Support/Attention

SUMMARY:
The purpose of this study is to compare three treatments to determine which is most effective in reducing anxiety in children.

DETAILED DESCRIPTION:
Children and their parents will complete a comprehensive diagnostic assessment to determine eligibility. The assessment will include an individual diagnostic interview with the child, interviews with the parents, and written observations of the child from family members and teachers. Participants will then be randomly assigned to receive individual cognitive behavioral therapy (ICBT), family CBT (FCBT), or education/support/attention (ESA) for 5 months. Children in the ICBT group will meet individually with a therapist. In the FCBT and ESA treatment groups, children and their parents will meet weekly with a therapist.

At the end of treatment and 1 year following treatment completion, families will complete another assessment to determine the effectiveness of each treatment at reducing short- and long-term anxiety symptoms in their children.

ELIGIBILITY:
Inclusion Criteria:

* Child with DSM-IV criteria for separation anxiety disorder, social phobia, or generalized anxiety disorder

Exclusion Criteria for Child Participants:

* IQ less than 80
* Current use of anti-anxiety or antidepressant medications
* Psychotic symptoms
* Child and/or parent is non-English speaking

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 2000-07

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Child and Adolescent Anxiety Disorders Clinic, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Kendall PC. Treating anxiety disorders in children: results of a randomized clinical trial. J Consult Clin Psychol. 1994 Feb;62(1):100-10. doi: 10.1037//0022-006x.62.1.100. PMID 8034812
- [Background] Kendall PC, Flannery-Schroeder E, Panichelli-Mindel SM, Southam-Gerow M, Henin A, Warman M. Therapy for youths with anxiety disorders: a second randomized clinical trial. J Consult Clin Psychol. 1997 Jun;65(3):366-80. doi: 10.1037//0022-006x.65.3.366. PMID 9170760